CLINICAL TRIAL: NCT03349307
Title: Feasibility of the Thin Convex Probe Endobronchial Ultrasound (TCP-EBUS) System for Lymph Node Staging
Brief Title: Thin-EBUS in Ex-vivo Human Lungs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-6083
Record Dates: First submitted 2017-11-13; First posted 2017-11-21 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Lung Cancer
Keywords: lobectomy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No Intervention (Experimental)
  Interventions: Device: Thin Convex Probe Endobronchial Ultrasound (TCP-EBUS)

INTERVENTIONS:
Device: Thin Convex Probe Endobronchial Ultrasound (TCP-EBUS) — Patients scheduled for a lobectomy will be recruited to this study and approached for informed consent. At the time of surgery, once the lobe has been removed, the TCP-EBUS will be inserted through a bronchial stamp for brief operability evaluations and image acquisition. Once this data has been captured standard of care will continue.

SUMMARY:
This study will determine the feasibility of the novel thin convex probe endobronchial ultrasound (TCP-EBUS) in human resected lobes. The primary end point is to clarify the feasibility of using the thin convex probe EBUS scope to visualize lung tumors from an intra-bronchial view. The secondary objective is to evaluate the insertion ability, operability, endoscopic image and ultrasound image compared to that of the convex probe EBUS.

ELIGIBILITY:
Inclusion Criteria:

* Any patients scheduled for lobectomy or anatomical segmental resection for malignant lung tumors.
* 18 years of age or older

Exclusion Criteria:

* Any patients with inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
To clarify the feasibility of using the thin convex probe EBUS scope to visualize lung tumors from an intra bronchial view. | Within an hour of resection.
  The TCP-EBUS bronchoscope will be inserted through the endotracheal tube for visualization of lobar, segmental and sub segmental bronchi.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The investigators plan to share data at the time of manuscript publication.